CLINICAL TRIAL: NCT03144141
Title: Association Between Holter Electro Hysterogram (EHG) and Risk of Preterm Delivery in Women Hospitalized for Threatened Premature Delivery
Brief Title: Association Between EHG and Risk of Preterm Delivery in Women Hospitalized for Threatened Premature Delivery
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0011
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with the diagnosis of threat of uterine delivery (Other)
  Interventions: Other: Electrical recording of uterine activity by EHG either directly at the emergency or at the hospitalization

INTERVENTIONS:
Other: Electrical recording of uterine activity by EHG either directly at the emergency or at the hospitalization — Electrical recording of uterine activity by EHG either directly at the emergency or at the hospitalization

SUMMARY:
Preterm delivery accounts for about 10% of deliveries in France. Prematurity is the leading cause of perinatal morbidity and mortality in economically developed countries. Despite the development of therapeutics and paraclinic examinations, this rate of preterm delivery remains stable or even increases. The use of medically assisted procreation techniques alone can not explain this rate.

The analysis of the electrical activity of the uterus (electrohysterograms) is a promising technique for early diagnosis of the risk of premature delivery, allowing better management of the patients. This study is part of a European theme to study risk factors for the prevention of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Patients arriving at maternity emergency for threat of premature birth between 26 SA and 35 SA defined by uterine contractions and a cervical modification
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient minor,
* Associated Obstetric Pathology: Pre-Eclampsia, Premature Rupture of Membranes (RPM)
* Patient under tutelage or curatorship or deprived of public law

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Analysis of the electrical activity of the uterus (electro hysterogram) for the early diagnosis of the risk of preterm delivery | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Result] https://theses.fr/2019COMP2489 Évaluation de l'électrohystérogramme pour la surveillance et le diagnostic des femmes à risque d'accouchement prématuré